CLINICAL TRIAL: NCT07142876
Title: Evaluation Of Liver Resection Using Harmonic Scalpel Versus Cavitron Ultrasonic Surgical Aspirator (CUSA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Mohamed Elzeer, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-8-5MD
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Liver Resection; Liver Tumours; Liver Transplant Disorder; Trauma Abdomen
Keywords: liver resection; CUSA; Cavitron Ultrasonic Surgical Aspirator; Harmonic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Abdominal Injuries | interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: prospective randomized comparative clinical trial study analyzing outcomes of liver resection by two different techniques CUSA or Harmonic scalpel .This will be a prospective comparative study at Sohag University Hospital and Assuit University Hospital, Egypt The study population was divided into two equal groups (25 per group) according to the method of liver transection: group A by CUSA and group B by harmonic scalpel (HS).
  Inclusion criteria patients needing liver resection in normal liver and cirrhotic liver child-pough A and early B with: Age > 6 and < 70 years old, One or two small (5 cm or less) hepatic lesions confined to the liver with no extra hepatic involvement, Patients with -ve markers for viral hepatitis.
  The exclusion criteria:
  patients with age < 6 or > 70 years old, liver cirrhosis Child-pough C, liver cell failure, very large lesions including most of the liver tissue, vascular invasion, evidence of metastasis in cases with HCC, positive hepatitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver resection with Cavitron Ultrasonic Surgical Settings Aspirator (CUSA) (Active Comparator): In-group A Cavitron Ultrasonic Surgical Settings Aspirator (CUSA) with standard tip was used for parenchymal transection with the following Settings; 23 kHz, 70 Watt, and continuous irrigation at rate of 4-6 ml/min with normal saline and the vessel coagulation was performed by the bipolar sealer (Valleylab force FX electrosurgical generator, Medtronic, Minneapolis, USA), the power was used at 50 Watt coagulation.
  Interventions: Procedure: Liver resection Cavitron Ultrasonic Surgical Aspirator (CUSA)
- Liver resection with the harmonic scalpel (Active Comparator): In group B the harmonic scalpel (Ethicon EndoSurgery, Johnson & Johnson, New Jersey, USA) was set at a high power, and blood vessels or bile ducts up to 3-4 mm in diameter were coagulated for 5-6 seconds.
  Interventions: Procedure: Liver resection with the harmonic scalpel

INTERVENTIONS:
Procedure: Liver resection Cavitron Ultrasonic Surgical Aspirator (CUSA) — In-group A Cavitron Ultrasonic Surgical Settings Aspirator (CUSA) with standard tip was used for parenchymal transection with the following Settings; 23 kHz, 70 Watt, and continuous irrigation at rate of 4-6 ml/min with normal saline and the vessel coagulation was performed by the bipolar sealer (Valleylab force FX electrosurgical generator, Medtronic, Minneapolis, USA), the power was used at 50 Watt coagulation.
  Other Names: Group A
  Arms: Liver resection with Cavitron Ultrasonic Surgical Settings Aspirator (CUSA)
Procedure: Liver resection with the harmonic scalpel — In group B the harmonic scalpel (Ethicon EndoSurgery, Johnson & Johnson, New Jersey, USA) was set at a high power, and blood vessels or bile ducts up to 3-4 mm in diameter were coagulated for 5-6 seconds.
  Other Names: Group B
  Arms: Liver resection with the harmonic scalpel

SUMMARY:
Evaluation Of Liver Resection Using Harmonic Scalpel Versus Cavitron Ultrasonic Surgical Aspirator (CUSA)

Introduction The mode of parenchymal transection in hepatic resection has been a topic of great debate for decades. Many resections have now evolved into laparoscopic , and robotic-assisted procedures to limit morbidity. Morbidity and mortality after hepatic resection has progressively improved over the years due to improved equipment, operative technique [3], and anesthetic management. Prior to 1980, mortality rates were reported to be in the 10-20% range with many deaths related to perioperative hemorrhage. Now perioperative mortality has dropped significantly to approximately 5%.

The clamp-crush technique, first reported in 1974, has been used for decades and remains the standard means of parenchymal division for many surgeons. Control of intraoperative hemorrhage has been one of the principle technical problems in advancing liver surgery. Excess blood loss and intraoperative blood transfusions have been shown to be associated with increased perioperative mortality and morbidity including an increased rate of hepatocellular carcinoma recurrence . Transfusions are also associated with increased infections and with increased cost. Costs of blood transfusions were recently examined in surgical patients.

Many devices are now available to surgeons for division of the liver parenchyma in both open and minimally invasive surgery including: the CUSA (Tyco Healthcare, Mansfield, MA), Harmonic Scalpel (Ethicon Endo-Surgery, Cincinnati, OH, USA), Ligasure (Valley Lab, Tyco Healthcare, Boulder, CO, USA), Tissue Link (Salient Surgical Technologies, Portsmouth, NH), water-jet dissection, radiofrequency, microwave assisted resection, vascular staplers, and others In this study, we looked at the TissueLink bipolar sealer device that was used in combination with the CUSA in group 1 termed the CUSA/TissueLink group, and the Harmonic Scalpel in the group 2 termed Harmonic Scalpel/TissueLink. The TissueLink uses radiofrequency energy focused near the end of the device for electrocautery and a low volume saline drip that produces ohmic heat causing precoagulation of hepatic parenchyma. The saline keeps the temperature at or below 100 C to avoid eshcar formation ultimately helping prevent delayed biliary leak and hemorrhage. The hemostatic effects of TissueLink are a result of its disruption of the collagen in blood vessels causing closing of the lumen .

The CUSA, a commonly used device in hepatic resection, was used in combination with the TissueLink in this study. We previously described this combination of devices reporting a shorter length of hospital stay, decreased operative time, and decreased intraoperative blood transfusion . CUSA uses ultrasonic energy to fragment and aspirate parenchymal tissue. This exposes biliary as well as vascular structures that may then be closed in a variety of ways at the surgeon's discretion. It allows for a precise transection plane allowing preservation of normal hepatic tissue .

The Harmonic Scalpel, used in this study in combination with the TissueLink, utilizes ultrasonic vibration of two blades causing destruction of hydrogen bonds. This disruption of hydrogen bonds causes protein denaturization coagulating small vessels of 3 mm diameter. The parenchyma is also cut when the blades move in a saw-like fashion In this study, we evaluated the safety and efficacy of two different techniques described above for the division of the hepatic parenchyma in order to improve perioperative outcomes.

DETAILED DESCRIPTION:
Evaluation Of Liver Resection Using Harmonic Scalpel Versus Cavitron Ultrasonic Surgical Aspirator (CUSA)

Introduction The mode of parenchymal transection in hepatic resection has been a topic of great debate for decades. Many resections have now evolved into laparoscopic , and robotic-assisted procedures to limit morbidity. Morbidity and mortality after hepatic resection has progressively improved over the years due to improved equipment, operative technique [3], and anesthetic management. Prior to 1980, mortality rates were reported to be in the 10-20% range with many deaths related to perioperative hemorrhage. Now perioperative mortality has dropped significantly to approximately 5%.

The clamp-crush technique, first reported in 1974, has been used for decades and remains the standard means of parenchymal division for many surgeons. Control of intraoperative hemorrhage has been one of the principle technical problems in advancing liver surgery. Excess blood loss and intraoperative blood transfusions have been shown to be associated with increased perioperative mortality and morbidity including an increased rate of hepatocellular carcinoma recurrence . Transfusions are also associated with increased infections and with increased cost. Costs of blood transfusions were recently examined in surgical patients.

Many devices are now available to surgeons for division of the liver parenchyma in both open and minimally invasive surgery including: the CUSA (Tyco Healthcare, Mansfield, MA), Harmonic Scalpel (Ethicon Endo-Surgery, Cincinnati, OH, USA), Ligasure (Valley Lab, Tyco Healthcare, Boulder, CO, USA), Tissue Link (Salient Surgical Technologies, Portsmouth, NH), water-jet dissection, radiofrequency, microwave assisted resection, vascular staplers, and others In this study, we looked at the TissueLink bipolar sealer device that was used in combination with the CUSA in group 1 termed the CUSA/TissueLink group, and the Harmonic Scalpel in the group 2 termed Harmonic Scalpel/TissueLink. The TissueLink uses radiofrequency energy focused near the end of the device for electrocautery and a low volume saline drip that produces ohmic heat causing precoagulation of hepatic parenchyma. The saline keeps the temperature at or below 100 C to avoid eshcar formation ultimately helping prevent delayed biliary leak and hemorrhage. The hemostatic effects of TissueLink are a result of its disruption of the collagen in blood vessels causing closing of the lumen .

The CUSA, a commonly used device in hepatic resection, was used in combination with the TissueLink in this study. We previously described this combination of devices reporting a shorter length of hospital stay, decreased operative time, and decreased intraoperative blood transfusion . CUSA uses ultrasonic energy to fragment and aspirate parenchymal tissue. This exposes biliary as well as vascular structures that may then be closed in a variety of ways at the surgeon's discretion. It allows for a precise transection plane allowing preservation of normal hepatic tissue .

The Harmonic Scalpel, used in this study in combination with the TissueLink, utilizes ultrasonic vibration of two blades causing destruction of hydrogen bonds. This disruption of hydrogen bonds causes protein denaturization coagulating small vessels of 3 mm diameter. The parenchyma is also cut when the blades move in a saw-like fashion In this study, we evaluated the safety and efficacy of two different techniques described above for the division of the hepatic parenchyma in order to improve perioperative outcomes.

Aim Of the Work This study was conducted aiming to assess the efficacy and safety of liver resection using Harmonic Scalpel Versus cavitron Ultrasonic Surgical Aspirator (CUSA)

Patients and methods The study design: prospective randomized comparative clinical trial study analyzing outcomes of liver resection by two different techniques CUSA or Harmonic scalpel .This will be a prospective comparative study at Sohag University Hospital and Assuit University Hospital, Egypt The study population was divided into two equal groups (25 per group) according to the method of liver transection: group A by CUSA and group B by harmonic scalpel (HS).

Inclusion criteria patients needing liver resection in normal liver and cirrhotic liver child-pough A and early B with: Age > 6 and < 70 years old, One or two small (5 cm or less) hepatic lesions confined to the liver with no extra hepatic involvement, Patients with -ve markers for viral hepatitis.

The exclusion criteria:

patients with age < 6 or > 70 years old, liver cirrhosis Child-pough C, liver cell failure, very large lesions including most of the liver tissue, hepatic lesions with vascular invasion, evidence of metastasis in cases with HCC, and patients with +ve markers for viral hepatitis.

Approvals and consents This study will be done after obtaining approval from the research ethics committee of the Sohag faculty of medicine. A written Informed consent will be obtained from all participants before being enrolled in the study and before performing the procedure after receiving an explanation of the study protocol, including both types of operation and possible complications.

The study will be registered at www.clinicaltrials.gov.

Data collection:

Registered data will be collected from the hospital databases, clinical data. Setting This study will be performed in Sohag University Hospital and Assuit University Hospital.

All operations will be performed under general anesthesia.

Preoperative:

All Patients underwent the following: Complete history taking and clinical examination focusing on: presenting symptoms, symptoms of chronic liver diseases (chronic hepatitis, liver cirrhosis) and jaundice, history of any preceding disease or previous operations and history of travelling to endemic areas. Laboratory investigation: Complete blood picture, Liver function tests: Albumin, bilirubin, ALT, AST, Coagulation profile, Renal function tests and Tumor markers: Alpha fetoprotein (AFP), CEA, and CA 19-9. Radiological evaluation: Abdominal ultrasound and Tri-phasic CT with hepatic venography, arteriography, portography and magnetic resonance cholangiopancreatography (MRCP) and residual liver volume must be more than or equals to 35%. ERCP: was performed in patients presented clinically with jaundice.

Surgical technique:

The procedure was performed through a right inverted J-shaped incision. Following laparotomy, liver mobilization and piggyback were done in the standard technique then an intra-operative ultrasound and cholangiogram were done to define the major biliary system anatomy and vasculature.

Transection of the liver parenchyma started from the anterocaudal liver surface toward the hepatic veins. The line of parenchymal transection was mapped about 1 cm to the right of the middle hepatic vein (MHV) using intraoperative Doppler ultrasound. The clearly exposed vessels (More than 5mm) were ligated by 4/0 or 5/0 polyprolene or clipped with preservation of V5 and V8.

In-group A Cavitron Ultrasonic Surgical Settings Aspirator (CUSA) with standard tip was used for parenchymal transection with the following Settings; 23 kHz, 70 Watt, and continuous irrigation at rate of 4-6 ml/min with normal saline and the vessel coagulation was performed by the bipolar sealer (Valleylab force FX electrosurgical generator, Medtronic, Minneapolis, USA), the power was used at 50 Watt coagulation.

In group B the harmonic scalpel (Ethicon EndoSurgery, Johnson & Johnson, New Jersey, USA) was set at a high power, and blood vessels or bile ducts up to 3-4 mm in diameter were coagulated for 5-6 seconds.

Following completion cholangiogram, open-suction silicon drain was placed into the subphrenic and subhepatic spaces close to the cut surface of the liver before abdominal wound closure.

Blood loss during parenchymal transection and immediately after hepatectomy until completion of the procedures was included and estimated by the volume of blood suctioned and subtraction of rinse fluids and/or weighting the swabs that were used during transection, (Every 1 mL of blood is equivalent to 1 g increase in the swab weight).

Postoperative bile leakage was diagnosed once bile was detected from the wound or the drain or drained intra-abdominal collection with total bilirubin level in the fluid more than 3 times that in the serum.

The liver resection time was defined as the duration from the beginning of parenchymal transection until the completion of transection with complete achievement of haemostasis from the liver cut surface.

Post-operative management All patients were admitted to the ICU for early post-operative care. Post-operative parameters of hepatic recovery, including serum total bilirubin, ALT, AST, prothrombin time, albumin, was measured daily until discharge from ICU then every other day till discharge.

The drain was removed when the amount drained was less than 100 mL/day and no bile leak and discharge from the hospital was based on the patient's general condition, clinical parameters, complications and abdominal ultrasound.

Follow-Up Upon discharge, all patients were followed once weekly with abdominal ultrasound together with routine laboratory data for at least 1 month.

ELIGIBILITY:
Inclusion Criteria:

* patients needing liver resection in normal liver and cirrhotic liver child-pough A and early B
* Age > 6 and < 70 years old
* One or two small (5 cm or less) hepatic lesions confined to the liver with no extra hepatic involvement
* Patients with -ve markers for viral hepatitis

Exclusion Criteria:

* patients with age < 6 or > 70 years old
* liver cirrhosis Child-pough C
* liver cell failure
* very large lesions including most of the liver tissue
* hepatic lesions with vascular invasion
* evidence of metastasis in cases with HCC
* patients with +ve markers for viral hepatitis

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative bile leakage | Day 14
  Postoperative bile leakage was diagnosed once bile was detected from the wound or the drain or drained intra-abdominal collection with total bilirubin level in the fluid more than 3 times that in the serum.
The liver resection time | Day 1
  The liver resection time was defined as the duration from the beginning of parenchymal transection until the completion of transection with complete achievement of haemostasis from the liver cut surface.
Blood loss | Day 1
  Blood loss during parenchymal transection and immediately after hepatectomy until completion of the procedures was included and estimated by the volume of blood suctioned and subtraction of rinse fluids and/or weighting the swabs that were used during transection, (Every 1 mL of blood is equivalent to 1 g increase in the swab weight).

SECONDARY OUTCOMES:
liver functions | Day 14
  Post-operative parameters of hepatic recovery, including serum total bilirubin, ALT, AST, prothrombin time, albumin, was measured daily until discharge from ICU then every other day till discharge.

CONTACTS AND LOCATIONS:
Overall Officials: AbdElaal A Prof. AbdElaal Ali Sleem, professor, Study Chair — AbdElaal Ali Sleem

IPD SHARING:
Plan to Share IPD: No
protecting my patients privacy and confidentiality